CLINICAL TRIAL: NCT01781676
Title: Registry Study Intensive Hospital Monitoring Protocol of Kudiezi Injection ( Yueanxin ) 's Clinical Safety
Brief Title: Safety Study of Kudiezi(Yueanxin,a Chinese Medicine Injection)Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, China Academy of Chinese Medical Sciences
Other Study IDs: RSCMI-Ⅷ
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Heart Disease; Angina Pectoris; Stroke
MeSH Terms: conditions — Coronary Disease; Angina Pectoris; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study was advocated by institute of Basic Research in Clinical Medicine,China Academy of Chinese Medical Sciences in October 2011.

It was funded by China major scientific and technological specialized specialized project for 'significant new formulation of net drugs'.

Kudiezi(Yueanxin) is kind of Chinese Medicine injiection used for treating corinary heart diswese、angina pectoris and stroke in many Chinese hospitals.

The purpose of this study is to determine adverse drug events or adverse drug reaction in large sample size 30,000 patients.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China.However safety problems rose in recent years.There could be many uncertain factors influence Chinese Medincine Injection in clinical practice.

Safety surveillance on Chinese Medincine injection is an important problem that needs to be sorted out through large sample observational dtudy.

A registry study for Kudiezi(Yueanxin) injection safety surveillance with 30000 patients will be conducted form Jan.2012 to Dec.2015.

Eligiblity crteria Patients who will use Kudiezi(Yueanxin) injection in selected hospitals.

Date will be collected in four aspects by four different forms as following:

Form A(blue):demographic information ;Form B(yellow):adverde drug events/reaction;Form C(white):extracted information from hodpiral information system and laboratory information system.

ELIGIBILITY:
Inclusion Criteria:

Patients using Kudiezi(Yueanxin) injection from 2012 to 2014

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticpcipated sample size was caculated in this study,about 30000.Patients using Kudiezi injection from 2012 to 2014 in more than 20 hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events;incidence of Kudiezi(Yueanxin)'ADRs and identify factors that contributed to the occurrence of the adverse reaction | to assess Kudiezi(Yueanxin)'s 'adverse event' and 'drug adverse reaction' during patients' hospital stay,administration information of Kudiezi will be registered every day.The registry procedure will last 3 years only for patients using Kudiezi.
  All patients will be measured and assessed at the time Kudiezi(Yueanxin) is adminnistered to them until they discharge.Patients using Kudiezi(Yueanxin) will be registered on a regisration form including disease background, Kudiezi(Yueanxin)'s adminidtration,and extraction information from hospital information system.An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients.A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Kudiezi(Yueanxin).

CONTACTS AND LOCATIONS:
Overall Officials: Xie Y Ming, BA, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Institute of Basic Research in Clinical Medicine, Beijing, Beijing Municipality, China